CLINICAL TRIAL: NCT00865098
Title: Open-label, Non-randomized, Non-controlled, Multicenter Phase II Study Investigating Cetuximab in Combination With Concomitant-boost Radiotherapy as First-line Treatment for Japanese Patients With Newly Diagnosed Locally Advanced SCCHN.
Brief Title: Study of Cetuximab With Concomitant-boost Radiotherapy in Patients With Newly Diagnosed Locally Advanced Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Yoshiteru Kimura, Merck Serono Co., Ltd. Tokyo, Japan, an Affiliate of Merck KGaA, Darmstadt, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 62241-053
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Results first posted 2011-07-22 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-02

CONDITIONS: Carcinoma of the Head and Neck
Keywords: Newly diagnosed locally advanced squamous cell carcinoma of the head and neck (SCCHN)
MeSH Terms: interventions — Cetuximab

ARMS (1):
- Cetuximab With Radiotherapy (Experimental)
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — Patients receive Cetuximab at an initial dose of 400 mg/m^2 of Cetuximab to be infused 6 or 7 days before starting radiotherapy, followed by subsequent weekly infusions at a dose of 250 mg/m^2 of Cetuximab and RT (72.0 Gy total in 42 fractions) for the next 6 weeks of the treatment course. Subjects will receive Cetuximab until radiographically documented progressive disease or unacceptable toxicity occurs or consent is withdrawn. If RT is delayed, administration of Cetuximab every 7 days is continued. If RT is discontinued for any reason, treatment with Cetuximab monotherapy every 7 days is continued.

SUMMARY:
This study is conducted in Japanese newly diagnosed locally advanced SCCHN patients in order to assess tolerability and feasibility of Cetuximab plus concomitant boost radiotherapy (RT) regimen (the study treatment) and its safety profile (i.e. AEs: adverse events). In addition, efficacy (i.e. anti-tumor effect) of the study treatment is also evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has pathologically proven squamous cell carcinoma arising in the oropharynx, hypopharynx, or larynx.
2. The patient has been confirmed Epidermal Growth Factor Receptor expressing in tumor specimen by immunohistochemistry.
3. The patient has stage III or IV disease (Unio Internationalis Contra Cancrum / International Union against Cancer Tumor-Lymph Nodes-Metastases classification) with an expected survival of ≥ 12 months.
4. The patient has at least bi-dimensionally measurable disease.
5. The patient is medically suitable to withstand a course of the definitive radiation therapy.
6. The patient aged ≥ 20 years old at informed consent
7. The patient's Karnofsky performance status is ≥ 60
8. Hemoglobin ≥ 9g/dL
9. Neutrophil ≥ 1500/mm^3
10. Platelet ≥ 100,000/mm^3
11. Total Bilirubin ≤ 1.5 mg/dL
12. Aspartate Aminotransferase ≤ 2 x the upper limit of normal
13. Alanine Aminotransferase ≤ 2 x the upper limit of normal
14. Serum creatinine ≤ 1.5 mg/dL
15. Serum calcium concentration: within normality
16. The patient is eligible if disease free from a previously treated malignancy for greater than three years.
17. The patient agrees to use effective contraception if procreative potential exists.
18. The patient has given signed informed consent
19. The patient who is a Japanese with Japanese citizenship

Exclusion Criteria:

1. The patient has evidence of distant metastatic disease. The patient who has any metastatic disease documented by Magnetic Resonance Imaging for the head and neck, and Computed Tomography for the chest and abdomen should be excluded.
2. The patient has squamous cell carcinoma arising in the nasopharynx or oral cavity.
3. The patient has received prior systemic chemotherapy within the last three years.
4. The patient has undergone previous surgery for the tumor under study other than biopsy.
5. The patient has received prior radiation therapy to the head and neck.
6. The patient's radiation therapy is considered to be a part of a postoperative regimen following primary surgical resection.
7. The patient is pregnant or breast feeding.
8. The patient has received prior Cetuximab or murine monoclonal antibody (including chimeric antibody) therapy or a history of severe hypersensitivity to any component of Cetuximab solution for Injection.
9. The patient has a medical or psychological condition that would not permit the patient to complete the study or sign informed consent (including drug abuse).
10. The patient has uncontrolled diabetes mellitus, malignant hypertension, or liver failure.
11. The patient has or has suffered from a pulmonary fibrosis, acute pulmonary disorder, or interstitial pneumonia.
12. The patient has an active infection (infection requiring intravenous anti-bacterial, anti-fungus, or anti-viral agent), or known and declared Human Immunodeficiency Virus infection.
13. The patient has a clinically relevant coronary artery disease or history of myocardial infarction in the last 12 months or high risk of uncontrolled arrhythmia or uncontrolled cardiac insufficiency
14. The patient has a dental disease which requires incision and drainage.
15. The patient has active multiple cancers (excluding skin cancer except for melanoma, and carcinoma in situ of the cervix or the digestive tract) in the last 3 years.
16. The patient has been received some investigational medication within 30 days before study entry.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masataka Ota, MD, Study Director — Merck Serono Co.,Ltd, an Affilate of Merck Serono, Darmstadt, Germany
Locations (4):
- Japan (4):
  - Research Site, Aichi
  - Research Site, Chiba
  - Research Site, Shizuoka
  - Research Site, Tokyo

REFERENCES:
- [Result] Okano S, Yoshino T, Fujii M, Onozawa Y, Kodaira T, Fujii H, Akimoto T, Ishikura S, Oguchi M, Zenda S, de Blas B, Tahara M, Beier F. Phase II study of cetuximab plus concomitant boost radiotherapy in Japanese patients with locally advanced squamous cell carcinoma of the head and neck. Jpn J Clin Oncol. 2013 May;43(5):476-82. doi: 10.1093/jjco/hyt030. Epub 2013 Mar 10. PMID 23479383

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in this study at 4 centers in Japan. The first subject was enrolled on 06 March 2009 and the last on 04 January 2010.
Pre-assignment Details: 27 subjects were enrolled and 5 were ineligible, not treated, and excluded from the Intention To Treat (ITT)/Safety Population. Reasons: investigator's decision (1 subject), withdrawal of consent (1 subject), inability to perform radiation therapy according to protocol (2 subjects) and inclusion/exclusion criteria not fulfilled (1 subject).
Groups:
- Cetuximab With Radiotherapy: Subjects received cetuximab at an initial dose of 400 mg/m² infused 6 or 7 days before starting radiotherapy (RT). This was followed by subsequent weekly infusions of 250 mg/m² cetuximab administered in combination with radiotherapy (5 days/week) for 6 weeks. Subjects will receive cetuximab until radiographically documented progressive disease or unacceptable toxicity occurs or consent is withdrawn. If RT is delayed, administration of cetuximab every 7 days is continued. If RT is discontinued for any reason, treatment with cetuximab monotherapy every 7 days is continued.
Period: Overall Study
Arm/Group | Cetuximab With Radiotherapy
Started | 22
Completed | 21 (Discontinued from the study due to progressive disease, after completing planned treatment schedule)
Not Completed | 1
Not completed — Progressive disease | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab With Radiotherapy
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (6.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 21
Region of Enrollment [Number; unit: participants]
  Japan | 22

OUTCOME MEASURES:

1. Primary Outcome: Completion Rate
Description: Number of subjects who complete ≥70% of Cetuximab planned dose administration in terms of relative dose intensity of Cetuximab and full dose of RT ≤2 weeks over planned schedule in terms of RT duration ≤8 weeks, divided by the the number of subjects in the ITT/Safety population
Time Frame: time from first administration of cetuximab to last administration of cetuximab or RT (whichever is later), ≤ 9 weeks
Population: ITT/Safety population, i.e. all subjects who have received at least one dose of the study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab With Radiotherapy
Number analyzed (Participants) | 22
percentage of participants | 100 [84.6 to 100.0]

2. Secondary Outcome: Best Response Rate
Description: Number of subjects experiencing a Complete Response (complete disappearance of measurable and evaluable disease without new lesions) or Partial Response (>=50% decrease of the sum of the product diameters of measurable disease, evaluable disease not worsening or progressing, no new lesions) at 8 weeks post radiotherapy (confirmed by repeat assessment at week 12) based on imaging according to modified World Health Organisation criteria as assessed independently by the Efficacy and Safety Evaluation Committee, divided by the number of subjects in the ITT/safety population
Time Frame: best response was determined at week 8 post radiotherapy, for subjects with complete or partial response a confirmation in week 12 post radiotherapy was required
Population: ITT/Safety population, i.e. all subjects who have received at least one dose of the study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab With Radiotherapy
Number analyzed (Participants) | 22
percentage of participants | 81.8 [59.7 to 94.8]

3. Secondary Outcome: Safety - Number of Patients Experiencing Any Adverse Event
Description: Please refer to Adverse Events section for further details
Time Frame: time from first dose up to 60 days after last dose of study treatment, ≤18 weeks
Population: ITT/Safety population, i.e. all subjects who have received at least one dose of the study treatment
Measure: Number; unit: participants
Arm/Group | Cetuximab With Radiotherapy
Number analyzed (Participants) | 22
participants | 22

4. Secondary Outcome: Safety - Number of Patients Experiencing Any Grade 4 Adverse Event
Description: Severity was assessed according to the toxicity criteria defined in the National Cancer Institute - Common Terminology Criteria for Adverse Event (NCI-CTCAE), Version 3.0, where grade 1 denoted mild, grade 2 moderate, grade 3 severe, and grade 4 lifethreatening or disabling. In the case of adverse events not contained within the NCI-CTCAE, the investigator was responsible for assessing the severity of the AE (grades 1 to 4) based on the jeopardy to the subject's health and well-being, and the ability of the subject to function during the event.
Time Frame: time from first dose up to 60 days after last dose of study treatment, ≤18 weeks
Population: ITT/Safety population, i.e. all subjects who have received at least one dose of the study treatment
Measure: Number; unit: participants
Arm/Group | Cetuximab With Radiotherapy
Number analyzed (Participants) | 22
participants | 2

5. Secondary Outcome: Safety - Number of Patients Experiencing Any Grade 3 or 4 Skin Reaction
Description: Skin reactions were considered as adverse events of special interest and were evaluated in a special AE category composed of specific MedDRA preferred terms. Severity was assessed according to criteria defined in the NCI-CTCAE, Version 3.0, where grade 1 is mild, grade 2 moderate, grade 3 severe, and grade 4 lifethreatening or disabling.
Time Frame: time from first dose up to 60 days after last dose of study treatment, ≤18 weeks
Population: ITT/Safety population, i.e. all subjects who have received at least one dose of the study treatment
Measure: Number; unit: participants
Arm/Group | Cetuximab With Radiotherapy
Number analyzed (Participants) | 22
participants | 3

6. Secondary Outcome: Safety - Number of Patients Experiencing Any Grade 3 or 4 Infusion Related Reaction
Description: Infusion related reactions were considered as adverse events of special interest and were evaluated in a special AE category composed of specific MedDRA preferred terms. Severity was assessed according to criteria defined in the NCI-CTCAE, Version 3.0, where grade 1 is mild, grade 2 moderate, grade 3 severe, and grade 4 lifethreatening or disabling.
Time Frame: time from first dose up to 60 days after last dose of study treatment, ≤18 weeks
Population: ITT/Safety population, i.e. all subjects who have received at least one dose of the study treatment
Measure: Number; unit: participants
Arm/Group | Cetuximab With Radiotherapy
Number analyzed (Participants) | 22
participants | 0

ADVERSE EVENTS:
Time Frame: Time from first dose up to 60 days after the last dose of study treatment. Adverse Events (AEs) are summarized using the MedDRA version 13.0.
Description: Treatment emergent Adverse Events (TEAEs) were defined as AEs that emerge or worsen on or after the first dosing day of trial treatment until 60 days after the last trial treatment administration.
Arm/Group | Cetuximab With Radiotherapy
Serious Adverse Events (participants affected / at risk) | 3/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab With Radiotherapy (N=22)
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Altered state of consciousness (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab With Radiotherapy (N=22)
Anaemia (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 2
Cheilitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 15
Diarrhoea (Gastrointestinal disorders) | 10
Dry mouth (Gastrointestinal disorders) | 17
Dyspepsia (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 4
Odynophagia (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 4
Mucosal inflammation (General disorders) | 19
Pyrexia (General disorders) | 11
Infection (Infections and infestations) | 5
Paronychia (Infections and infestations) | 5
Pharyngitis (Infections and infestations) | 2
Radiation skin injury (Injury, poisoning and procedural complications) | 10
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 2
Blood albumin decreased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 2
Blood urea increased (Investigations) | 2
Weight decreased (Investigations) | 9
Decreased appetite (Metabolism and nutrition disorders) | 10
Dehydration (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 5
Hyponatraemia (Metabolism and nutrition disorders) | 2
Dysgeusia (Nervous system disorders) | 15
Headache (Nervous system disorders) | 2
Delirium (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 3
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 14
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 11
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 8
Dry skin (Skin and subcutaneous tissue disorders) | 15
Pruritus (Skin and subcutaneous tissue disorders) | 10
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Skin fissures (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other